CLINICAL TRIAL: NCT04813250
Title: The Effects of Ventilatory Strategies on Pulmonary Function After Cardiopulmonary Bypass Evaluated by Electrical Impedance Tomography in Patients Undergoing Cardiac Surgery
Brief Title: Ventilatory Strategies After Cardiopulmonary Bypass Evaluated by Electrical Impedance Tomography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Defense Medical Center, Taiwan (Other)
Responsible Party: Principal Investigator, Yung-Chi Hsu, Attending Physician of Department of Anesthesiology, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Ventilatory with EIT post CPB
Record Dates: First submitted 2021-03-21; First posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Elective Cardiac Surgical Patients
Keywords: Ventilatory strategies; Electrical Impedance Tomography; cardiac surgery

STUDY DESIGN:
Intervention Model Description: Ventilation strategies with 4 different ventilation mode since weaning cardiopulmonary bypass (CPB), Four group were control EtCO2 between 35～45mmHg by adjusting respiratory rate, EIT Measurements were performed under supine position
Who Masked: Outcomes Assessor
Masking Description: De-identify the data before analyse the data by outcome saaessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group R (Sham Comparator): IMV(intermittent mandatory ventilation) Regular Ventilation with Tidal volume with 7ml/ kg (Predicted body weight)
  Interventions: Other: ventilation mode setting
- Group RP (Experimental): Regular Ventilation with Tidal volume with 7ml/ kg (Predicted body weight) + PEEP : 6 cm H2O
  Interventions: Other: ventilation mode setting
- Group RI (Experimental): Regular Ventilation with Tidal volume with 7ml/ kg (Predicted body weight) + Reverse IE ratio ventilation( I:E=1:1)
  Interventions: Other: ventilation mode setting
- Group RPI (Experimental): Regular Ventilation with Tidal volume with 7ml/ kg (Predicted body weight) + PEEP : 6 cm H2O + Reverse IE ratio ventilation( I:E=1:1)
  Interventions: Other: ventilation mode setting

INTERVENTIONS:
Other: ventilation mode setting — Ventilation strategies with 4 kinds of ventilator mode since weaning cardiopulmonary bypass (CPB), Four group were control EtCO2 between 35～45mmHg by adjusting respiratory rate, EIT Measurements were performed under supine position

SUMMARY:
Pulmonary complications after cardiac surgeries are common. It is one of the most crucial concerns of cardiac surgeons and anesthesiologists. These adverse events may vary from a mild respiratory dysfunction to acute respiratory distress syndrome (ARDS). One of the most public reasons of these complications is atelectasis that would result in hypoxia and pneumonia. Any of these adverse events rises the prevalence of morbidity and mortality. The chief inducing causes for atelectasis are CPB and dropped blood perfusion and ventilation of the lungs. The ventilation arrest is related with a high frequency of retained bronchial sections, local atelectasis, decrease in arterial O2 concentrations as a effect of surge in arteriovenous shunt, declined lung compliance, pulmonary edema and hence increased risk of nosocomial infections.

Electrical Impedance Tomography (EIT) is a non-invasive, radiation-free, real time bedside imaging modality, which provide the assessment of regional gas volume and lung ventilation. EIT has been experienced in quite a lot of animal and clinical applications including optimization of mechanical ventilator strategies and recognition of respiratory adverse events. Besides, EIT has been used to recognize ideal PEEP by detection of homogenous ventilation in non-dependent and dependent lung regions. Homogeneous ventilation is key for inhibition of ventilator-induced lung injury.

DETAILED DESCRIPTION:
The aim of this study is to use four different ventilatory strategies 【Group R : IMV(intermittent mandatory ventilation) Regular Ventilation with Tidal volume with 7ml/ kg (Predicted body weight) ； Group RP, Regular Ventilation with Tidal volume with 7ml/ kg (Predicted body weight) + PEEP : 6 cm H2O ；Group RI : Regular Ventilation with Tidal volume with 7ml/ kg (Predicted body weight) + Reverse IE ratio ventilation( I:E=1:1) ；Group RPI: Regular Ventilation with Tidal volume with 7ml/ kg (Predicted body weight) + PEEP : 6 cm H2O + Reverse IE ratio ventilation( I:E=1:1)】 to compare the beneficial in decreasing the incidence of post-operative pulmonary dysfunction after cardiac surgery including of the data of EIT, GAS , Lactate , PFR：PaO2/FiO2 ratio , cardiac index (CI) , BMI..etc . EIT were measured at two perioperative timepoints 1. after intubation at the onset of anesthesia with mechanical ventilation with 7ml/ kg (Predicted body weight) 2. at the end of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-80 year-old
* Adult patients receiving elective cardiac surgery with hypothermic CPB

Exclusion Criteria:

* Patients were excluded if they had complicating comorbidities, such as chronic hepatic or renal insufficiency, acute cardiopulmonary failure requiring mechanical ventilation, intra-aortic balloon pump, or extracorporeal membrane oxygenation

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
The correlation between Different ventilation mode and the relevant value of EIT | since weaning cardiopulmonary bypass (CPB) to the end of surgery
  Compare the correlation between Different ventilation mode and the relevant value of EIT in the population of open heart surgery patient
The demographic characteristics and relevant value of EIT | since weaning cardiopulmonary bypass (CPB) to the end of surgery
  Campare the demographic characteristics and relevant value of EIT in the population of open heart surgery patient

SECONDARY OUTCOMES:
If the different ventilation mode setting can improve clinical outcome | since weaning cardiopulmonary bypass (CPB) to the end of surgery
  Identify the different ventilation mode setting in open heart surgery patient if can improve clinical care benifit.
The correlation between heart function & oxygenation and different ventilation mode | since weaning cardiopulmonary bypass (CPB) to the end of surgery
  Survey the correlation between heart function & oxygenation and different ventilation mode

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, Tri-Service General Hospital, Taipei, Neihu Dist, Taiwan

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Spinelli E, Mauri T, Fogagnolo A, Scaramuzzo G, Rundo A, Grieco DL, Grasselli G, Volta CA, Spadaro S. Electrical impedance tomography in perioperative medicine: careful respiratory monitoring for tailored interventions. BMC Anesthesiol. 2019 Aug 7;19(1):140. doi: 10.1186/s12871-019-0814-7. PMID 31390977